CLINICAL TRIAL: NCT00587418
Title: L-arginine Supplement for the Prevention of Calcineurin Inhibitor Nephrotoxicity
Brief Title: L-arginine for Prevention of Kidney Damage in Liver Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, W. Ray Kim, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-007047; R21AT004174 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Liver Transplant Recipients
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arginine (Experimental)
  Interventions: Dietary Supplement: L-arginine
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine — Arginaid (Novartis) 1 package (9.2g) bid for 7 days
  Arms: Arginine
Dietary Supplement: Placebo — Placebo powder 9.2g bid for 7 days
  Arms: Placebo

SUMMARY:
Chronic renal insufficiency is a common and important health problem that causes morbidity and mortality among patients who have undergone liver transplantation. It is mainly caused by drugs (calcineurin inhibitors) that are used to prevent or treat rejection and once established, there is no effective treatment. This research investigates whether L-arginine can reverse the effects of calcineurin inhibitors on the kidneys and thus prevent renal insufficiency in liver transplant recipients.

DETAILED DESCRIPTION:
Although liver transplantation (LTx) is now well-established as a means of restoring health in patients with liver failure, there remain opportunities to further optimize its outcome. One of the major sources of mortality and morbidity in LTx recipients is renal insufficiency associated with nephrotoxicity of immunosuppressant agents, particularly calcineurin inhibitors (i.e., cyclosporine and tacrolimus). These agents are also associated with hypertension and diabetes among LTx recipients, contributing to further reduction in renal function. In a report based on nationwide data, 18% of LTx recipients developed renal failure within 5 years.

Most of the decline in renal function after LTx occurs in the first few months. This is in part because patients are exposed to the highest levels of calcineurin inhibitors in the early post-LTx period, when the risk of acute cellular rejection is the greatest. Calcineurin inhibitors produce intense renal vasoconstriction, which may be reversible early on. Over time, however, irreversible changes, such as vascular angiopathy, tubular atrophy and eventually interstitial fibrosis, contribute to permanent reduction in renal perfusion and glomerular filtration. Thus, interventions to preserve renal function after LTx would be most effective in the early post-LTx period, when most reduction in renal function occurs and when renal vascular changes are potentially reversible.

Existing evidence and our preliminary data indicate that impairment of vasodilatory response mediated by nitric oxide (NO) plays an important role in the pathogenesis of calcineurin inhibitor nephrotoxicity. Our overall hypothesis is that L-arginine supplement provides protection against calcineurin inhibitor nephrotoxicity. L-arginine, a naturally occurring amino acid, is the main substrate of the NO synthase enzyme and exogenous supplementation of L-arginine may improve renal perfusion by inducing renal vasodilation via increased NO production. Although L-arginine has been shown to prevent renal damage from calcineurin inhibitors in experimental animals, its efficacy in preserving renal function has not been studied in human LTx recipients.

In this application, we propose to conduct a pilot, randomized, double-blinded, placebo-controlled trial to explore the use of prophylactic L-arginine supplement in preserving renal function in LTx recipients. Twenty-four (24) LTx recipients recovering uneventfully from the procedure will be recruited for the study. Subjects will be randomized 1:1 to receive 9g per day of L-arginine or placebo given orally for 7 days between 14 and 21 days after LTx, followed by open-label maintenance with L-arginine. The aims of the study are as follows:

AIM 1. To determine the effect of oral L-arginine supplement on glomerular filtration rate in LTx recipients. We will compare changes in GFR, as estimated by the eGFRcys equation, before and after a 7-day trial of L-arginine versus placebo. The eGFRcys equation has recently been shown to be the most accurate GFR estimator incorporating serum cystatin-C and creatinine concentrations, age, gender and race.

AIM 2. To determine the effect of L-arginine supplement on secondary efficacy endpoints. We will compare plasma L-arginine concentrations and urinary cyclic-GMP, the latter being a key metabolite of renal NO, between the L-arginine and placebo groups.

AIM 3. To evaluate the safety of oral L-arginine supplement in liver transplant recipients. We will compare the frequency and severity of adverse events between the L-arginine and placebo groups.

AIM 4. To determine the effect of maintenance open label L-arginine on GFR. After the 7-day trial, participants will be offered an open label L-arginine for 13 additional weeks. We will compare their GFR determined by iothalamate clearance before and after the maintenance use of L-arginine supplement.

Our hypothesis is that L-arginine will promote the release of NO in the renal vascular bed, increasing renal blood flow and glomerular filtration rate (AIM 1). We believe it is critical that we test this in patients early after LTx before irreversible vascular and glomerular damage is established. Once this proof of concept is attained, we would like to link the observation with plasma L-arginine concentration and urinary c-GMP excretion (AIM 2). Based on extensive experience at Mayo Clinic of using oral L-arginine, we expect to demonstrate no clinically significant adverse events with L-arginine (AIM 3). The data from the open label maintenance phase (AIM 4) will help gauge whether the short term benefit shown in AIM 1 is sustainable for a longer time frame.

The significance of these studies is based on several factors: (1) Calcineurin inhibitor-induced renal insufficiency is a major source of morbidity and mortality among LTx recipients; (2) Once it is established, there is no effective treatment for calcineurin inhibitor-induced renal insufficiency; and (3) If the results of this study support our hypothesis, we will be able to embark upon a full scale, randomized trial of long-term oral L-arginine supplement using GFR as the end point. Such a study will be able to answer whether a simple amino acid supplement may prevent calcineurin inhibitor nephrotoxicity, making a fundamental difference in morbidity, mortality and quality of life of our patients, who have undergone a life-changing procedure, namely liver transplantation.

ELIGIBILITY:
Inclusion criteria

1. Informed written consent
2. Ages 18+ at the time of entry into the study
3. Recipient of primary liver transplantation from a deceased or live donor
4. Stable with satisfactory allograft function

   1. Total bilirubin < 2.5 mg/dl and
   2. Aminotransferase < x 3 upper limit of normal (e.g., ALT<120 IU/mL)
5. Serum creatinine < 2.5 mg/dl without dialysis
6. Maintenance immunosuppression including tacrolimus or cyclosporine
7. Stable hemodynamic function

   1. Systolic blood pressure > 100 mmHg
   2. Resting pulse rate < 100

Exclusion criteria

1. Recipient of combined liver-kidney transplantation
2. Prior organ transplantation (i.e., exposure to calcineurin inhibitors)
3. Established primary renal disease with active urinary sediments
4. On-going renal replacement therapy
5. Pulmonary hypertension (e.g., portopulmonary hypertension)
6. Iodine allergy
7. Other systemic illness (e.g., infection) that require hospitalization care beyond 2 weeks after LTx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes in eGFR before and after L-arginine | 7 days with option for 12 week maintenance phase

SECONDARY OUTCOMES:
Urinary excretion of cGMP before and after L-arginine. Creatinine before and after L-arginine. | 7 days with option for 12 week maintenance phase
Safety of oral L-arginine | 7 days with option for 12 week maintenance phase
Change in iothalamate clearance before and after optional 12 week maintenance open label phase. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: W. Ray Kim, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States